CLINICAL TRIAL: NCT05999383
Title: Understanding the Clinical Pharmacology of Marijuana-Tobacco Co-administration
Acronym: CANNIC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institutes of Health (NIH) (NIH); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 23-38884; 1R01DA056451-01A1 (NIH)
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: THC; Cannabis; Cannabis Use; Cannabis Smoking; Tobacco Use; Vaping
Keywords: THC; Cannabis; Marijuana; Nicotine; Vape
MeSH Terms: conditions — Marijuana Abuse; Marijuana Smoking; Tobacco Use; Vaping | interventions — nabiximols; Nicotine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Placebo marijuana and regular cigarette (Experimental): Participants will vape a 50/50 mixture of placebo marijuana (0% THC) and regular cigarette (25.94 mg/g nicotine content)
  Interventions: Drug: Nicotine; Device: Pax Loose Leaf Vaporizer; Other: Placebo Marijuana
- Placebo marijuana and Very Low Nicotine Content cigarette (Experimental): Participants will vape a 50/50 mixture of placebo marijuana (0% THC) and Very Low Nicotine Content cigarette (0.42 mg/g nicotine content)
  Interventions: Drug: Nicotine; Device: Pax Loose Leaf Vaporizer; Other: Placebo Marijuana
- Medium marijuana and regular cigarette (Experimental): Participants will vape a 50/50 mixture of medium marijuana (<5% THC) and regular cigarette (25.94 mg/g nicotine content)
  Interventions: Drug: Cannabis; Drug: Nicotine; Device: Pax Loose Leaf Vaporizer
- Medium marijuana and Very Low Nicotine Content cigarette (Experimental): Participants will vape a 50/50 mixture of medium marijuana (<5% THC) and Very Low Nicotine Content cigarette (0.42 mg/g nicotine content)
  Interventions: Drug: Cannabis; Drug: Nicotine; Device: Pax Loose Leaf Vaporizer
- High marijuana and regular cigarette (Experimental): Participants will vape a 50/50 mixture of high marijuana (>10% THC) and regular cigarette (25.94 mg/g nicotine content)
  Interventions: Drug: Cannabis; Drug: Nicotine; Device: Pax Loose Leaf Vaporizer
- High marijuana and Very Low Nicotine Content cigarette (Experimental): Participants will vape a 50/50 mixture of high marijuana (>10% THC) and Very Low Nicotine Content cigarette (0.42 mg/g nicotine content)
  Interventions: Drug: Cannabis; Drug: Nicotine; Device: Pax Loose Leaf Vaporizer
- High marijuana only (Experimental): Participants will vape high marijuana (>10% THC)
  Interventions: Drug: Cannabis; Device: Pax Loose Leaf Vaporizer
- Regular cigarette only (Experimental): Participants will vape a regular cigarette (25.94 mg/g nicotine content)
  Interventions: Drug: Nicotine; Device: Pax Loose Leaf Vaporizer

INTERVENTIONS:
Drug: Cannabis — Participants will vape marijuana in varying doses from the PAX device
  Other Names: Marijuana
  Arms: High marijuana and Very Low Nicotine Content cigarette; High marijuana and regular cigarette; High marijuana only; Medium marijuana and Very Low Nicotine Content cigarette; Medium marijuana and regular cigarette
Drug: Nicotine — Participants will vape Regular and Very Low Nicotine content cigarettes from the PAX device
  Other Names: Nicotine product
  Arms: High marijuana and Very Low Nicotine Content cigarette; High marijuana and regular cigarette; Medium marijuana and Very Low Nicotine Content cigarette; Medium marijuana and regular cigarette; Placebo marijuana and Very Low Nicotine Content cigarette; Placebo marijuana and regular cigarette; Regular cigarette only
Device: Pax Loose Leaf Vaporizer — In all arms, participants will be using the PAX Loose Leave Vaporizer.
  Other Names: Electronic vaporizor
Other: Placebo Marijuana — Participants will vape placebo marijuana from the PAX device
  Other Names: Placebo for Marijuana
  Arms: Placebo marijuana and Very Low Nicotine Content cigarette; Placebo marijuana and regular cigarette

SUMMARY:
This is a crossover, randomized, double-blinded clinical pharmacology study enrolling dual cannabis-tobacco smokers to better understand the combined effects of co-administering cannabis and tobacco. The project aims to describe the pharmacokinetics and pharmacodynamics of marijuana-tobacco co-administration by delivering THC and nicotine in various combinations. This foundational study will establish a research program focused on elucidating the public health consequences of marijuana-tobacco co-use.

DETAILED DESCRIPTION:
This is a single-center, within-subject (crossover), randomized, double-blinded clinical pharmacology study of over 8 study visits (days). Participants will be non-treatment-seeking, healthy frequent users of both marijuana and tobacco/nicotine, age 21 to 65 years (21 years because of California tobacco control law). Participants will be marijuana users of any race who smoke or vape marijuana or THC extracts at least three days a week for the past 3 months or more. The study investigators will use positive urine toxicology THC results and self-report of marijuana smoking/vaping to determine eligibility. Participants must also be current users of inhaled forms of tobacco/nicotine (cigarettes, cigars, e-cigarettes) who use the product daily over the past 3 months.

Each study day will consist of a standardized session of 5 puffs of one of 8 study conditions using a PAX-3 vaporizer (PAX Labs, Inc.). Blood will be sampled multiple times for plasma THC, nicotine, and catecholamines, questionnaires administered for sensory and subjective effects, and heart rate, skin blood flow, and skin temperature will be measured. After 6 hours of abstinence, participants will have 60 minutes of ad libitum access to the assigned study condition, during which heart rate and blood pressure will be continuously monitored, blood sampled before and after for THC, nicotine, and platelet aggregation measured, and questionnaires administered.

Studies will be conducted at the Clinical & Translational Science Institute (CTSI) Clinical Research Services-supported research ward at Zuckerberg San Francisco General.

ELIGIBILITY:
Inclusion Criteria:

* Heart rate < 105 beats per minute (BPM)*
* Systolic Blood Pressure < 160 and > 90*
* Diastolic Blood Pressure < 100 and > 50*

  *Considered out of range if both machine and manual readings are above/below these thresholds.
* Body Mass Index (BMI) ≤ 38.0 (at investigator's discretion for higher BMI if no other concurrent health issues)
* Current regular user of cannabis who smokes or vapes cannabis or THC extracts at least three days a week for the past 3 months or more
* Test positive for D-9-tetrahydrocannabinol (THC) at screening and self-report of cannabis use
* Current user of inhaled forms of tobacco/nicotine (cigarette, cigars, e-cigarettes) who use the product daily for the past 3 months or more
* Saliva cotinine ≥ 30 ng/mL

Exclusion Criteria:

* Unstable medical conditions:

  * Heart disease
  * Seizures
  * Cancer
  * Thyroid disease (okay if controlled with medication)
  * Diabetes
  * Hepatitis B or C or Liver disease
  * Glaucoma
  * Kidney disease or urinary retention
  * An ulcer in the past year
  * Active use of an inhaler for asthma or Chronic Obstructive Pulmonary Disease (COPD)
* Hypertension if uncontrolled (meaning participant has a diagnosis, but they are not taking medication/under treatment (e.g., diet or exercise plan)
* Drug/Alcohol Dependence

  * Alcohol or illicit drug dependence within the past 12 months (currently in treatment) with the exception of those who recently completed an alcohol/drug treatment program
  * Positive toxicology test at the screening visit (THC & prescribed medications okay)
  * Opioid replacement therapy (including methadone, buprenorphine, or other)
* Psychiatric conditions

  * Current or past schizophrenia, and/or current or past bipolar disorder
  * Major depression, current or within the past year
  * Major personality disorder
  * Participants with current or past minor or moderate depression and/or anxiety disorders will be reviewed by the PI [study physician] and considered for inclusion
  * History of psychiatric hospitalizations are not exclusionary, but study participation will be determined as per PI's [study physician's] approval
* Current regular use of any psychiatric medications with the exception of Selective serotonin reuptake inhibitors (SSRI) and serotonin-norepinephrine reuptake inhibitors (SNRI) and current evaluation by the PI that the participant is otherwise healthy, stable, and able to participate
* Congenital or acquired immunodeficiency disorders (i.e. HIV, congenital immune deficiency syndrome, chronic diseases)
* Other disorders (i.e. ICU, malnutrition, immunosuppressive therapy)
* Traumatic brain injury
* Recent onset or change (worsening) in cough, fever and/or abdominal symptoms (vomiting or pain) in the past two weeks
* Medications

  * Use of medications that are inducers of nicotine metabolizing enzyme CYP2A6 (Example: rifampicin, dexamethasone, phenobarbital, and other anticonvulsant drugs)
  * Concurrent use of nicotine-containing medications
  * Any stimulant medications (ex. Adderall) generally given for attention deficit hyperactivity disorder (ADHD) treatment
* Other/Misc. Chronic Health Problems

  * Oral thrush
  * Fainting
  * Other "life threatening illnesses" as per study physician's discretion
* Pregnancy

  * Pregnancy (self-reported and urine pregnancy test)
  * Breastfeeding (determined by self-report)
* Concurrent participation in another clinical trial
* Inability to communicate in English
* History of marijuana-induced psychosis or paranoia after smoking marijuana
* Scoring a 7 or higher on the Severity of Dependence Scale (SDS) for cannabis use
* Planning to quit smoking or vaping within the next 60 days
* Planning to quit cannabis use within the next 60 days
* Uncomfortable with getting blood drawn
* Willingness to abstain from tobacco smoking and all combustible products for 13 hours before admission
* Willingness to abstain from smoking/ingestion of cannabis 13 hours before
* Willingness to abstain from nicotine products 13 hours before each admission

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in peak plasma concentration of THC | From Baseline to Day 1
  To assess the differences between THC dosages, the study investigators will determine maximum plasma THC concentration (Cmax) using plasma THC concentrations from the standardized sessions.
Change in peak plasma concentration of THC | From Day 1 to Day 2
  To assess the differences between THC dosages, the study investigators will determine maximum plasma THC concentration (Cmax) using plasma THC concentrations from the standardized sessions.
Change in peak plasma concentration of THC | From Day 2 to Day 3
  To assess the differences between THC dosages, the study investigators will determine maximum plasma THC concentration (Cmax) using plasma THC concentrations from the standardized sessions.
Change in peak plasma concentration of THC | From Day 3 to Day 4
  To assess the differences between THC dosages, the study investigators will determine maximum plasma THC concentration (Cmax) using plasma THC concentrations from the standardized sessions.
Change in peak plasma concentration of THC | From Day 4 to Day 5
  To assess the differences between THC dosages, the study investigators will determine maximum plasma THC concentration (Cmax) using plasma THC concentrations from the standardized sessions.
Change in peak plasma concentration of THC | From Day 5 to Day 6
  To assess the differences between THC dosages, the study investigators will determine maximum plasma THC concentration (Cmax) using plasma THC concentrations from the standardized sessions.
Change in peak plasma concentration of THC | From Day 6 to Day 7
  To assess the differences between THC dosages, the study investigators will determine maximum plasma THC concentration (Cmax) using plasma THC concentrations from the standardized sessions.
Change in peak plasma concentration of THC | From Day 7 to Day 8
  To assess the differences between THC dosages, the study investigators will determine maximum plasma THC concentration (Cmax) using plasma THC concentrations from the standardized sessions.
Change in Peak plasma concentration of nicotine | From Baseline to Day 1
  To assess the differences between nicotine dosages, the study investigators will determine maximum plasma nicotine concentration (Cmax) using plasma nicotine concentrations from the standardized sessions.
Change in Peak plasma concentration of nicotine | From Day 1 to Day 2
  To assess the differences between nicotine dosages, the study investigators will determine maximum plasma nicotine concentration (Cmax) using plasma nicotine concentrations from the standardized sessions.
Change in Peak plasma concentration of nicotine | From Day 2 to Day 3
  To assess the differences between nicotine dosages, the study investigators will determine maximum plasma nicotine concentration (Cmax) using plasma nicotine concentrations from the standardized sessions.
Change in Peak plasma concentration of nicotine | From Day 3 to Day 4
  To assess the differences between nicotine dosages, the study investigators will determine maximum plasma nicotine concentration (Cmax) using plasma nicotine concentrations from the standardized sessions.
Change in Peak plasma concentration of nicotine | From Day 4 to Day 5
  To assess the differences between nicotine dosages, the study investigators will determine maximum plasma nicotine concentration (Cmax) using plasma nicotine concentrations from the standardized sessions.
Change in Peak plasma concentration of nicotine | From Day 5 to Day 6
  To assess the differences between nicotine dosages, the study investigators will determine maximum plasma nicotine concentration (Cmax) using plasma nicotine concentrations from the standardized sessions.
Change in Peak plasma concentration of nicotine | From Day 6 to Day 7
  To assess the differences between nicotine dosages, the study investigators will determine maximum plasma nicotine concentration (Cmax) using plasma nicotine concentrations from the standardized sessions.
Change in Peak plasma concentration of nicotine | From Day 7 to Day 8
  To assess the differences between nicotine dosages, the study investigators will determine maximum plasma nicotine concentration (Cmax) using plasma nicotine concentrations from the standardized sessions.

SECONDARY OUTCOMES:
Cardiovascular effects among dosages using heart rate as a measure | From Baseline to Day 1
  The investigators will compare maximum change in heart rate as well as an integrated measure of heart rate over the first 180 minutes after the standardized session among dosages.
Cardiovascular effects among dosages using heart rate as a measure | From Day 1 to Day 2
  The investigators will compare maximum change in heart rate as well as an integrated measure of heart rate over the first 180 minutes after the standardized session among dosages.
Cardiovascular effects among dosages using heart rate as a measure | From Day 2 to Day 3
  The investigators will compare maximum change in heart rate as well as an integrated measure of heart rate over the first 180 minutes after the standardized session among dosages.
Cardiovascular effects among dosages using heart rate as a measure | From Day 3 to Day 4
  The investigators will compare maximum change in heart rate as well as an integrated measure of heart rate over the first 180 minutes after the standardized session among dosages.
Cardiovascular effects among dosages using heart rate as a measure | From Day 4 to Day 5
  The investigators will compare maximum change in heart rate as well as an integrated measure of heart rate over the first 180 minutes after the standardized session among dosages.
Cardiovascular effects among dosages using heart rate as a measure | From Day 5 to Day 6
  The investigators will compare maximum change in heart rate as well as an integrated measure of heart rate over the first 180 minutes after the standardized session among dosages.
Cardiovascular effects among dosages using heart rate as a measure | From Day 6 to Day 7
  The investigators will compare maximum change in heart rate as well as an integrated measure of heart rate over the first 180 minutes after the standardized session among dosages.
Cardiovascular effects among dosages using heart rate as a measure | From Day 7 to Day 8
  The investigators will compare maximum change in heart rate as well as an integrated measure of heart rate over the first 180 minutes after the standardized session among dosages.
Area under the plasma concentration versus time curve (AUC) | From Baseline to Day 1
  To assess the differences of absorption among dosages, the study investigators will determine the AUC using plasma nicotine and THC concentrations from the standardized sessions.
Area under the plasma concentration versus time curve (AUC) | From Day 1 to Day 2
  To assess the differences of absorption among dosages, the study investigators will determine the AUC using plasma nicotine and THC concentrations from the standardized sessions.
Area under the plasma concentration versus time curve (AUC) | From Day 2 to Day 3
  To assess the differences of absorption among dosages, the study investigators will determine the AUC using plasma nicotine and THC concentrations from the standardized sessions.
Area under the plasma concentration versus time curve (AUC) | From Day 3 to Day 4
  To assess the differences of absorption among dosages, the study investigators will determine the AUC using plasma nicotine and THC concentrations from the standardized sessions.
Area under the plasma concentration versus time curve (AUC) | From Day 4 to Day 5
  To assess the differences of absorption among dosages, the study investigators will determine the AUC using plasma nicotine and THC concentrations from the standardized sessions.
Area under the plasma concentration versus time curve (AUC) | From Day 5 to Day 6
  To assess the differences of absorption among dosages, the study investigators will determine the AUC using plasma nicotine and THC concentrations from the standardized sessions.
Area under the plasma concentration versus time curve (AUC) | From Day 6 to Day 7
  To assess the differences of absorption among dosages, the study investigators will determine the AUC using plasma nicotine and THC concentrations from the standardized sessions.
Area under the plasma concentration versus time curve (AUC) | From Day 7 to Day 8
  To assess the differences of absorption among dosages, the study investigators will determine the AUC using plasma nicotine and THC concentrations from the standardized sessions.
Change in subjective effects scores using the Marijuana Cravings Questionnaire (MCQ) | From Baseline to Day 1
  Self-assessed cravings will be measured using the MCQ. Questions on the MCQ are scored on a 7 point scale of 1 = Strongly Disagree and 7 = Strongly Disagree, with higher scores indicating increased cravings.
Change in subjective effects scores using the Marijuana Cravings Questionnaire (MCQ) | From Day 1 to Day 2
  Self-assessed cravings will be measured using the MCQ. Questions on the MCQ are scored on a 7 point scale of 1 = Strongly Disagree and 7 = Strongly Disagree, with higher scores indicating increased craving of marijuana.
Change in subjective effects scores using the Marijuana Cravings Questionnaire (MCQ) | From Day 2 to Day 3
  Self-assessed cravings will be measured using the MCQ. Questions on the MCQ are scored on a 7 point scale of 1 = Strongly Disagree and 7 = Strongly Disagree, with higher scores indicating increased cravings.
Change in subjective effects scores using the Marijuana Cravings Questionnaire (MCQ) | From Day 3 to Day 4
  Self-assessed cravings will be measured using the MCQ. Questions on the MCQ are scored on a 7 point scale of 1 = Strongly Disagree and 7 = Strongly Disagree, with higher scores indicating increased cravings.
Change in subjective effects scores using the Marijuana Cravings Questionnaire (MCQ) | From Day 4 to Day 5
  Self-assessed cravings will be measured using the MCQ. Questions on the MCQ are scored on a 7 point scale of 1 = Strongly Disagree and 7 = Strongly Disagree, with higher scores indicating increased cravings.
Change in subjective effects scores using the Marijuana Cravings Questionnaire (MCQ) | From Day 5 to Day 6
  Self-assessed cravings will be measured using the MCQ. Questions on the MCQ are scored on a 7 point scale of 1 = Strongly Disagree and 7 = Strongly Disagree, with higher scores indicating increased cravings.
Change in subjective effects scores using the Marijuana Cravings Questionnaire (MCQ) | From Day 6 to Day 7
  Self-assessed cravings will be measured using the MCQ. Questions on the MCQ are scored on a 7 point scale of 1 = Strongly Disagree and 7 = Strongly Disagree, with higher scores indicating increased cravings.
Change in subjective effects scores using the Marijuana Cravings Questionnaire (MCQ) | From Day 7 to Day 8
  Self-assessed cravings will be measured using the MCQ. Questions on the MCQ are scored on a 7 point scale of 1 = Strongly Disagree and 7 = Strongly Disagree, with higher scores indicating increased cravings.

CONTACTS AND LOCATIONS:
Overall Officials: Gideon St Helen, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No